CLINICAL TRIAL: NCT05786417
Title: A Trial Comparing the Effectiveness and Tolerability of Medications in Older Adults With Stable Angina and Multiple Chronic Conditions: LIVEBETTER
Brief Title: LIVEBETTER: A Trial Comparing Medications in Older Adults With Stable Angina and Multiple Chronic Conditions
Acronym: LIVEBETTER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000034470; HA-2021C3-24767 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI)); K76AG088428 (NIH)
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-02

CONDITIONS: Angina; Stable Ischemic Heart Disease
MeSH Terms: conditions — Angina Pectoris | interventions — Adrenergic beta-Antagonists; Calcium Channel Blockers

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized (1:1), 640 Older Adults with SIHD and MCC and 101 caregivers
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Beta-Blockers (BB) Therapy (Experimental): Participants randomized to this arm will be given a beta-blocker. Specific and appropriate drug selection from the class of beta blockers (i.e. type of BB, dosing, and escalation of dose) will be left to the site clinician in accordance with clinical guidelines. All BB will be administered orally (i.e. pills).
  Interventions: Other: Clinician Discretion; Drug: Beta blocker
- Calcium Channel Blockers (CCB) Therapy (Experimental): Participants randomized to this arm will be given a calcium channel blocker. Specific and appropriate drug selection from the class of calcium channel blockers (i.e. type of CCB, dosing, and escalation of dose) will be left to the site clinician in accordance with clinical guidelines. All CCB will be administered orally (i.e. pills).
  Interventions: Other: Clinician Discretion; Drug: Calcium channel blocker

INTERVENTIONS:
Other: Clinician Discretion — Clinician discretion as to which BB or CCB will be used if the participant has a heart rate and blood pressure within normal limits.
Drug: Beta blocker — Selection of the specific BB and initial starting dose will be determined by the treating clinician.
  Arms: Beta-Blockers (BB) Therapy
Drug: Calcium channel blocker — Selection of the specific CCB and initial starting dose will be determined by the treating clinician.
  Arms: Calcium Channel Blockers (CCB) Therapy

SUMMARY:
To establish the effectiveness and tolerability of standard of care anti-anginal treatment (beta-blocker and calcium channel blocker medications) in older adults with symptomatic Stable Ischemic Heart Disease (SIHD) and multiple chronic conditions (MCC).

DETAILED DESCRIPTION:
Single-blind, randomized (1:1) pragmatic trial comparing Beta-Blocker therapy versus Calcium Channel Blocker therapy in older adults with symptomatic SIHD and MCC with plans to initiate medical treatment with anti-anginal therapy.

Study Aims Aim 1: To compare the effectiveness of anti-anginal medications to improve the symptoms, function, and quality of life among older adults with multiple chronic conditions presenting with stable angina. Aim 2: To compare the tolerability and safety of commonly used anti-anginal medications in older adults with multiple chronic conditions presenting with stable angina. Aim 3 (Exploratory): To compare the long-term effectiveness and safety of specific anti-anginal medicine treatment approaches in older adults with multiple chronic conditions presenting with stable angina. LIVEBETTER consists of 4 study visits during the 12-month follow-up period. Visits are comprised of an interview, six-minute walk, and medical record review. Medication dose and administration will be addressed as part of routine clinical care.

The importance of the knowledge gained includes the following:

1. LIVEBETTER will produce randomized contemporary data on the safety and efficacy of BBs vs CCBs with the goal of filling that gap of evidence in the guidelines and informing clinical practice.
2. LIVEBETTER will generate data on the quality of life, symptomatic, and functional outcomes most pertinent to older adults with multiple chronic conditions and stable angina.
3. LIVEBETTER will provide the first quantitative data on caregiver burden in older adults with stable angina.

Cognition as measured by the Telephone Interview for Cognitive Status (TICS) is an exploratory endpoint included in the parent LIVEBETTER study. In November 2024, additional exploratory neurocognitive study measures were added as part of an ancillary neurocognitive study funded by the National Institute on Aging in September 2024. Additional measures introduced as part of this ancillary study include an extended cognitive battery and instruments to assess depression and functional status. As part of the ancillary neurocognitive study, study follow-up will be extended to 24 months. The exploratory aims of the neurocognitive ancillary study will be to compare the effect of BB vs. CCB on the rate of cognitive decline and incidence of mild cognitive impairment (MCI) and probable dementia among older adults with stable angina and MCC in the LIVEBETTER randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

OLDER ADULTS WITH SIHD AND MCC

* Age ≥65 years
* ≥ 2 Multiple Chronic Conditions as defined by Centers for Medicare and Medicaid Services (CMS)
* Diagnosis of Symptomatic Stable Ischemic Heart Disease with plans to initiate medical therapy identified by at least one of the following:

  1. positive non-invasive functional or anatomic testing suggestive of obstructive coronary artery disease
  2. coronary angiography with stenosis ≥70% in a coronary artery ≥2 mm in diameter or

     ≥50% stenosis of left main
  3. Invasive coronary angiography with positive physiologic testing in at least one vessel (FFR ≤ 0.80 or iFR ≤0.89)

CAREGIVERS

* Age ≥ 18 years
* Identified as caregiver of LIVEBETTER participant

Exclusion Criteria:

OLDER ADULTS WITH SIHD AND MCC

* Current taking (both) a beta-blocker AND a calcium channel blocker*
* Contraindication to beta-blockers or calcium channel blockers including:

  1. significant hypotension
  2. high grade AV block
  3. severe symptomatic bradycardia
  4. severe obstructive lung disease
* Documented intolerance to beta-blockers or calcium channel blockers
* Probable or definite high-risk coronary artery disease including unrevascularized left main disease and/or unrevascularized multi-vessel disease including the proximal left anterior descending (LAD) artery with plans for immediate complete revascularization
* Plans for complete revascularization within 2 weeks
* Clear clinical indication for beta-blockers or calcium channel blockers that precludes dose adjustment or crossover:

  1. Diagnosis of acute coronary syndrome (ACS) with reduced ejection fraction within past year
  2. Heart failure with reduced ejection fraction (HFrEF) within past year
* Actively participating in another clinical trial involving an investigational medication or device
* Primary language other than English or Spanish
* Inability to complete follow-up (e.g. life expectancy <12 months, impaired decision-making determined by validated instrument)
* Previously enrolled in LIVEBETTER
* Refused informed consent

CAREGIVERS

* Professional caregiver (i.e. not a relative or close friend of the participant)
* Primary language other than English or Spanish
* Inability to complete follow-up
* Previously enrolled in LIVEBETTER
* Refused informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 741 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life assessed using EQ-5D-5L | Baseline and 45 days
  The EQ-5D-5L represents a global quality of life measure that includes multiple components potentially impacted by the anti-anginal treatments being examined. The EQ-5D-5L score includes questions on mobility, self-care, usual activities, anxiety/depression, and pain/discomfort on a 5-point scale: 1=No Problem, 2=Slight Problem, 3=Moderate Problem, 4=Severe Problem, 5=Extreme Problem or Inability. 0, 1, and negative values corresponding to death, full health, and health states worse than death, respectively. Higher scores indicated greater levels of problems across each of the five dimensions.

SECONDARY OUTCOMES:
Change in Persistence on medication | up to 6 months
  Persistence on anti-anginal medication in the assigned treatment arm, as verified through a combination of the medical records (medication administration) and through self-report. Persistence is defined as either "Persistent" on treatment or "Not persistent" on treatment.
Change in Quality of Life assessed using EQ-5D-5L | Baseline, 6 months, 12 months, 24 months
  The EQ-5D-5L represents a global quality of life measure that includes multiple components potentially impacted by the anti-anginal treatments being examined. The EQ-5D-5L score includes questions on mobility, self-care, usual activities, anxiety/depression, and pain/discomfort on a 5-point scale: 1=No Problem, 2=Slight Problem, 3=Moderate Problem, 4=Severe Problem, 5=Extreme Problem or Inability. 0, 1, and negative values corresponding to death, full health, and health states worse than death, respectively. Higher scores indicated greater levels of problems across each of the five dimensions.
Change in Quality of Life assessed using PROMIS® Scale v1.2 - Global Health | Baseline, 45 days, 6 months, 12 months, 24 months
  The PROMIS Scale measures Physical Function (PF), Pain Interference (PI) and Anxiety Components with T - Score = 50 = General Population Mean.
  A Score > 50 = Better Physical Function, Less anxiety and decreased pain A Score < 50 = Poor Physical Function, More anxiety, and increased pain.
Change in Angina Control assessed using Seattle Angina Questionnaire (SAQ) Summary Score | Baseline, 45 days, 6 months, 12 months, 24 months
  The 7-item SAQ instrument captures the frequency of angina with the SAQ Angina Frequency score (and conversely "freedom from angina"), disease-specific effect of angina on physical function with the SAQ Physical Limitation score and quality of life with the Quality of Life score; these scores average to the SAQ Summary score. The scale of the score ranges from 0 - 100. 0 to 24 represents poor health status, 25 to 49 as fair, 50 to 74 as good, and 75 to 100 as excellent.
Change in 6-minute walk test | Baseline and 45 days
  The 6-minute walk test provides a more objective quantitative measure of mobility, functional performance, and symptom control. It measures the distance an individual can walk over a total of six minutes on a hard, flat surface. The individual can self-pace and rest as needed as they walk back and forth along a marked course. The participant can use an assistive walking device they normally use, such as a cane. The minimum clinically important difference in 6-minute walk distance is approximately 30 meters, a difference that is associated with mortality.
Change in Caregiver Burden Inventory | Baseline, 45 days, 6 months, 12 months, 24 months
  24-item questionnaire measuring caregiver burden with 5 subscales: (a) Time Dependence; (b) Developmental; (c) Behavior; (d) Physical Burden; (e) Social Burden; (f) Emotional Burden. This measure will provide insight into the degree to which treatment with different anti-anginal therapies impacts caregiver burden. Scores from subscales are summed for total score. The maximum score (maximum burden) is 96, with a minimum possible score of 0. A total score >36 indicates a risk of caregiver burnout whereas scores near or slightly >24 indicate a need to seek respite care.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nanna, MD, Principal Investigator — Yale University
Locations (9):
- United States (9):
  - Yale School of Medicine, New Haven, Connecticut
  - Wellstar Research Institute, Marietta, Georgia
  - Cook County Health, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mt. Sinai Health System, New York, New York
  - NYC Health and Hospitals, Harlem Hospital, New York, New York
  - Nirvana Integrative Medicine, New York, New York
  - Duke University, School of Medicine, Durham, North Carolina
  - Inova Health Care Services, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be available but de-identified and deposited into a Patient-Centered Outcomes Research Institute (PCORI)-endorsed repository when the study is complete.